CLINICAL TRIAL: NCT06490458
Title: Effects of Balance Training Post Coronary Artery Bypass Grafting
Brief Title: Effects of Balance Training on Functional Capacity of Patients After Coronary Artery Bypass Grafting Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Collaborators: National Heart Institute, Egypt (Other Government)
Responsible Party: Principal Investigator, Hady Atef Labib, Lecture of cardiopulmonary rehabilitation, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: balance and cabg patients
Record Dates: First submitted 2024-06-30; First posted 2024-07-08 (Actual); Last update posted 2024-07-08 (Actual); Status verified 2024-06

CONDITIONS: Coronary Artery Bypass Graft Surgery(CABG)
MeSH Terms: interventions — Cardiac Rehabilitation

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A :( Study group) (Active Comparator): Underwent balance training and cardiac rehabilitation program for a duration of 25-30 min (total session) at a frequency of three times/week (every other day). The balance training was: a- Functional strength exercise b- Stance exercise c- Transition exercise D-Gait training e- Cardiac rehabilitation program .
  Interventions: Combination Product: Balance Training
- Group B (control group) (Active Comparator): underwent cardiac rehabilitation program only for a duration of 25-30 min (total session) at a frequency of three times/week (day after day).
  the control group, received cardiac rehabilitation program only.
  Interventions: Combination Product: Balance Training

INTERVENTIONS:
Combination Product: Balance Training — Balance exercises and cardiac rehabilitation (intervention) for patients for 7 Days, 3 times/week for duration of 25-30 min/ session.
  Other Names: cardiac rehabilitation

SUMMARY:
Background:There are still many gaps in research concerning the effect of balance training on functional capacity of patient after coronary artery bypass graft.

Aims: The purpose of this study was to examine the effect of balance training on patients after coronanry artery bypass graft surgery.

DETAILED DESCRIPTION:
Methods: Sixty male patients under went CABG with ages 55-65 years Patients were randomly randomized into to two groups equal in number 30 in each group. (Group A: study group, Group B: control group).All patients were thoroughly evaluated one day after extubation and day 6 after operation.

Berg Balance Scale (BBS): is a test used to assess patients functional balance , the sit to stand test(STS) used to asses patients functional capacity and SF36 is questionnaire used to assess quality of life with patients. all of those tests done before and after training sessions with both groups. and compare the length of hospital stay between both groups.

ELIGIBILITY:
Inclusion Criteria:

1. Sixty male patients underwent CABG surgery, their age between 55 to 65 years old.
2. All patients were conscious, clinically and medically stable.
3. All patients are ambulant independently.
4. All patients are haemodynamically stable.
5. Good cognition level.
6. All patients are conscious and can perform physical activity.

Exclusion Criteria:

1. Hemodynamic instability.
2. Patients who need re-intubation.
3. Patients on high inotropic supports.
4. Patients with existing pulmonary disease or associated pulmonary complications.
5. Recent MI.
6. Patients who reported too much pain.
7. Neuromuscular disorders.
8. Active hemorrhage and hemoptysis.
9. Poor cognition and mentality.
10. Unstable angina.
11. Decompensated heart failure.
12. Deep vein thrombosis.

Ages: 55 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — male patients their age ranged from 55 to 65
Enrollment: 60 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2023-12-10 (Actual); Study Completion 2023-12-10 (Actual)

PRIMARY OUTCOMES:
Berg balance scale(BBS) | 7 Days
  (0 indicating the lowest level ,4 indicating the highest level ) data about balance from BBS index.

SECONDARY OUTCOMES:
sit to stand test(SST)in seconds | 1st day and 7th day
  represent functional capacity (duration of 5 times sit to stand)
length of hospital stay (in Days) | from 1st day
  number of days spent in hospital
SF36 Questionnaire( scores) | 3rd day
  Scores range from 0 - 100 Lower scores = more disability, higher scores = less disability

CONTACTS AND LOCATIONS:
Overall Officials: Hady Balabel, phD, Principal Investigator — Cairo University
Locations (1):
- National heart institute, Giza, Egypt

IPD SHARING:
Plan to Share IPD: Yes
after approval can be shared
Supporting Information: Study Protocol
Time Frame: after 1 month for 12 months
Access Criteria: will upload it to the journal of publication

REFERENCES:
- [Derived] Atef H, Marques-Sule E, Moreno-Segura N, Maged A, ELSayed SH, Pengelly J, Ali HF, Ghaffar HAE. Impact of early balance training on recovering following coronary artery bypass grafting. A randomized trial. Clin Rehabil. 2025 Dec 30:2692155251407320. doi: 10.1177/02692155251407320. Online ahead of print. PMID 41468033